CLINICAL TRIAL: NCT03582917
Title: The Role of VitD in Rehabilitation of Idiopathic Adolescent Scoliosis
Acronym: ScoliVit
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Assistant Professor of PMR, Orthopaedic Spine Surgeon, University of Ioannina
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UIoannina
Record Dates: First submitted 2018-05-29; First posted 2018-07-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alphacalscidol (Experimental): 0,5mg tablet by mouth, one each day for one year
  Interventions: Drug: Alphacalcidol
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Alphacalcidol — Alphacalcidol 0,5mg tablet
  Arms: Alphacalscidol

SUMMARY:
The purpose of this current prospective study is to determine the role of vitamin D in the development and restoration of spinal deformities in adolescence.

DETAILED DESCRIPTION:
The investigator will record the medical history of each patient and information such as age, body size (weight, height) and body mass index (BMI = kg / m ^ 2). Girls will also be given the time of appearance of menstruation, a factor that needs to be evaluated because the growth of the skeleton continues three years after its appearance. Patients will be subjected to Adam's Test, x-ray's and as well as lateral bending radiographs.In the first contact with each patient, will be evaluated bone density measured by DEXA as well as haematological testing including PTH, alkaline phosphatase (ALP), calcium (Ca), phosphorus( P ), Calcitonin and, of course, vitamin D (total and metabolite 25 (OH) D).

Each patient's follow-up will be completed in two years by a clinical examination every six months and a clinical, laboratory and radiological examination per year. Patients will be divided into two groups. In a group with patients with normal 25 (OH) D and in a second group with patients with low levels of 25 (OH) D. Members of the second group will receive substitution treatment with an appropriate formulation. The results will be collected and evaluated using statistical programme.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Adolescent Scoliosis
* Risser sign <3-4

Exclusion Criteria:

* Neuromuscular diseases
* metabolic disease
* Liver, lung, thyroid and parathyroid gland disorders.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Patients will be boys aged 10 to 18 and girls 10 to 16
Enrollment: 80 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
25(OH)D | 48 weeks
  Measurement of the major metabolite of vitamin D
X - rays | 48 weeks
  Cobb angle measurement
Dexa | 48 weeks
  BMD and Z - score measurement
BMD (weight in kilograms, height in meters) | 48 weeks
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (2):
- Greece (2):
  - Papanikolaou General Hospital, Asvestochóri
  - Department of Physical Medicine and Rehabilitation, University Hospital of Ioannina, Ioannina